CLINICAL TRIAL: NCT02729389
Title: The Effects of Experimentally Manipulated Social Status on Energy Balance in Youth: A Randomized Controlled Trial
Brief Title: Influence of Monopoly Game on Subtle Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Alabama at Birmingham (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201600361
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Psychosocial Influence on Cardiovascular Disease; Cardiovascular Disease
Keywords: Social Status; Hispanics; Energy Balance; Stress
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Social Status Condition (Experimental): Participants will be provided with a high degree of privilege in a game of Monopoly.
  Interventions: Behavioral: High Social Status Condition
- Low Social Status Condition (Experimental): Participants will be provided with a low degree of privilege in a game of Monopoly.
  Interventions: Behavioral: Low Social Status Condition

INTERVENTIONS:
Behavioral: High Social Status Condition — Participants will be provided with a high degree of privilege in a game of Monopoly.
  Arms: High Social Status Condition
Behavioral: Low Social Status Condition — Participants will be provided with a low degree of privilege in a game of Monopoly.
  Arms: Low Social Status Condition

SUMMARY:
The purpose of this research study is to investigate how social standing in a game of Monopoly may influence behavior.

DETAILED DESCRIPTION:
Participants will be asked to fill out questionnaires/surveys and health measures will be collected throughout the study visit. These health measures will include: blood pressure, heart rate, height/weight, waist circumference, percent body fat, resting metabolic rate, and salivary cortisol. Breakfast will be provided and then a 40-minute game of Monopoly™ will be played, and lunch will be provided after the game. Participants will be given an accelerometer to measure movements, and a food diary to be used for a 24-hour period. Once the 24-hour monitoring period has been completed, the participants will be finished with the study activities. The accelerometer and food diary will be returned by either bringing them to the investigators or mailing the items back to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic American adolescents born in the United States
* Have played Monopoly before

Exclusion Criteria:

* Clinical depression
* A diagnosis of cardiovascular disease (active or within the past 6 months), cancer (active or within the past 2 years, except non-melanoma skin cancer), diabetes (type 1 or 2), active or chronic infections, gastrointestinal disease, active kidney disease, lung disease, uncontrolled psychiatric disease
* An eating disorder or severely restricted diet
* Use of tobacco products
* Substance abuse disorder
* Take any medications known to affect appetite or body composition
* Participation in any weight-reduction programs, weight-loss diets, or other special diets within the previous 3 months
* Experience of weight loss or gain of 10 pounds or more of body weight in the past 6 months for any reason except post-partum weight loss
* Current/Anticipation of pregnancy during study
* Currently nursing or within 6 weeks of having completed nursing

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Energy balance between the groups at hour 4 and over 24 hours | Hour 4, After 24 Hours
  The investigators will assess energy balance using accelerometry, consumption data and resting metabolic rate.

SECONDARY OUTCOMES:
Change in blood pressure between the groups at hours 0, 1, 3, 4 | Hours 0, 1, 3, 4
  Systolic and diastolic blood pressure will be assessed.
Change in heart rate between the groups at hours 0, 1, 3, 4 | Hours 0, 1, 3, 4
  Heart rate will be captured using a heart rate monitor.
Change in salivary cortisol between the groups at hours 1, 3 | Hours 1, 3
  Salivary cortisol will be collected and tested to determine objective stress levels.
Change in Visual Analog Scales (VAS) between the groups at hours 0, 1, 3, 4 | Hours 0, 1, 3, 4
  Scores are from 0 - 100, 0 generally meaning least and 100 generally meaning most.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle I Cardel, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Translational Science Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee AM, Huo T, Miller D, Gurka MJ, Thompson LA, Modave FP, Hong YR, Pavela G, Cardel MI. The effects of experimentally manipulated social status and subjective social status on physical activity among Hispanic adolescents: An RCT. Pediatr Obes. 2022 May;17(5):e12877. doi: 10.1111/ijpo.12877. Epub 2021 Dec 3. PMID 34859604
- [Derived] Cardel MI, Pavela G, Janicke D, Huo T, Miller D, Lee AM, Gurka MJ, Dhurandhar E, Peters JC, Caldwell AE, Krause E, Fernandez A, Allison DB. Experimentally Manipulated Low Social Status and Food Insecurity Alter Eating Behavior Among Adolescents: A Randomized Controlled Trial. Obesity (Silver Spring). 2020 Nov;28(11):2010-2019. doi: 10.1002/oby.23002. PMID 33150744